CLINICAL TRIAL: NCT03832153
Title: Pan-Cardio-Genetics Clot Assessment in Acute Coronary Syndromes
Acronym: PGCA-ACS
Status: Withdrawn | Type: Observational
Why Stopped: LACK OF FUNDING
Sponsor: Aristotle University Of Thessaloniki (Other)
Collaborators: HELLENIC CENTER FOR MARINE RESEARCH (Unknown); Harvard Medical School (HMS and HSDM) (Other); Centre for Research and Technology Hellas (Other)
Responsible Party: Principal Investigator, Karagiannidis Efstratios, Medical Doctor (resident physician, Cardiology Department, AHEPA University hospital), PhD candidate, Principal Investigator, Aristotle University Of Thessaloniki
Other Study IDs: 20181028
Record Dates: First submitted 2019-01-27; First posted 2019-02-06 (Actual); Last update posted 2022-03-03 (Actual); Status verified 2022-02

CONDITIONS: STEMI - ST Elevation Myocardial Infarction; Thrombi; MicroRNA
Keywords: Bioprinting; thrombus aspiration; micro-CT
MeSH Terms: conditions — ST Elevation Myocardial Infarction; Thrombosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Intracoronary blood samples will be collected (during thrombus aspiration) along with peripheral blood samples and will be analyzed for the presence of specific micro-RNAs.
  The aspirated thrombi will be preserved in 10% formalin solution and will be analyzed using the Micro/Nano-CT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with low thrombus burden: patients with the lower volume of aspirated thrombi, as measured using micro-CT
  Interventions: Procedure: thrombus aspiration
- patients with high thrombus burden: patients with the higher volume of aspirated thrombi, as measured using micro-CT
  Interventions: Procedure: thrombus aspiration

INTERVENTIONS:
Procedure: thrombus aspiration — Thrombus aspiration will be performed by experienced interventional cardiologists according to standard practices, as previously described. The intracoronary blood samples will be collected as well during the same procedure and- along with peripheral blood samples- they will be analyzed for the presence of specific miRNAs. The aspirated thrombi will be preserved in 10% formalin solution and will be analyzed using the micro/nano-CT scanners.

SUMMARY:
Acute myocardial infarction with ST elevation (STEMI) is one of the leading causes of mortality. Although the presence of thrombus in STEMI patients has been linked to adverse outcomes, routine thrombus aspiration has not been proven effective. A potential explanation could be that patients with STEMI should be risk-stratified. Thus, a more personalized approach in treating these patients is stressfully required. This proposal aims to establish the required interdisciplinary infrastructure for developing a risk-stratification model by implementing clinical, laboratory and angiographic data with molecular knowledge obtained by using innovative technologies, such as data from nano/micro-Computed tomography and circulating microRNAs. Two hundred consecutive patients with STEMI undergoing thrombus aspiration will be enrolled in the study and will be followed-up for one year for Major Adverse Cardiac and Cerebrovascular events (MACCE). The proposed approach will shed light on the pathophysiological mechanisms and broaden the investigator's understanding of the complex cellular and molecular interactions in the STEMI setting that, along with clinical parameters, affect patient outcomes. Furthermore, it will enable the identification of certain circulating micro-RNAs as cardiovascular disease biomarkers and it will help clinicians to better stratify the cardiovascular and cerebrovascular risk of patients with STEMI. As part of the work, important characteristics of aspirated thrombi will be assessed for the first time (such as volume, density and shape) and will be linked to patient outcomes. All this information will be incorporated into one in-vitro model, which will be developed using bioprinting and microfluidics methodologies. The in-vitro model will facilitate: (i) the in-depth exploration of the pathophysiological mechanisms in patients with STEMI; and (ii) the therapeutic optimization of innovative nanocarriers/nanomedicines with thrombolytic efficacy. Clearly, the study improves personalized cardiovascular medicine approaches, by considering individual patient clinical assessment in a way that empowers the precision in diagnosis and therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptoms of myocardial ischemia lasting for more than 30 minutes
* Definite ECG changes indicating STEMI
* Patients undergoing primary PCI within 12 hours from symptom onset
* Possibility to perform thrombus aspiration
* Written informed consent

Exclusion Criteria:

* Treatment with fibrinolytic therapy for qualifying index STEMI event
* Patients with known intolerance to aspirin, ticagrelor or heparin
* Patients with active internal bleeding
* Patients with a recent history of intracranial hemorrhage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 210 consecutive patients presenting with STEMI and undergoing thrombus aspiration will be enrolled in the study
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2022-03-30 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
Fold changes of differentially-expressed microRNA from peripheral blood from patients suffering from STEMI (measured in log2 scale) | 12 months
  The expression profiles of the total number of microRNAs that exist in the peripheral blood of patients suffering from STEMI will be analyzed using Next Generation Sequencing (NGS). Blood samples collected from the patients will be used to extract microRNAs through the application of suitable microRNA isolation kit (miRNeasy Serum/Plasma kit). Following, the miRNA library construction will be prepared using commercially available reagents (QIAseq miRNA Library kit). The quantification of miRNAs will be done by the Qubit dsDNA HS assay kit in the Qubit fluorometer before the cDNA library generation.Statistical analyses of differentially expressed miRNAs will be carried out using EdgeR by the generalized linear model. Fold changes of differentially-expressed microRNA will be measured in log2 scale.
Volume of aspirated thrombus burden | 12 months
  The volume of aspirated thrombi will be quantified (in mm3) using micro-CT.

SECONDARY OUTCOMES:
Association between fold changes of microRNA expression and post-procedural Thrombolysis in Myocardial Infarction (TIMI) flow | 12 months
  Fold changes of differentially-expressed microRNAs (measured in log2 scale as described above) will be correlated to post-procedural TIMI flow (classified as previously described: TIMI flow 0,1,2 or 3).
Association between fold changes of microRNA expression (measured in log2 scale) with distal embolization | 12 months
  Fold changes of differentially-expressed microRNAs (measured in log2 scale, as described above) will be correlated to distal embolization (dichotomous variable-yes/no).
Association between fold changes of microRNAs expression and volume of aspirated thrombus. | 12 months
  Fold changes of differentially-expressed microRNA (measured in log2 scale) will be correlated to the volume of aspirated thrombi (measured in mm3), as it will be quantified using micro-CT.
Association between fold changes of microRNA expression and Major Adverse Cardiovascular and Cerebrovascular Events (MACCE) | 12 months
  Fold changes of differentially-expressed microRNAs (measured in log2 scale) will be correlated to MACCE. MACCE are defined as any of the following: cardiac death, cerebrovascular death, acute myocardial infarction, target lesion revascularization, stent thrombosis or stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Sianos, Study Chair — Associate Professor of Cardiology, Aristotle University of Thessaloniki; Ioannis Vizirianakis, Principal Investigator — Associate Professor, School of Pharmacy, Aristotle University of Thessaloniki; Dimitrios Fatouros, Principal Investigator — Associate Professor in Pharmaceutical Technology , Aristotle University of Thessaloniki; Eleftherios Angelis, Principal Investigator — Professor in Statistics, Aristotle University of Thessaloniki; Christos Arvanitidis, Principal Investigator — Director of Research, Hellenic Center for Marine Research; James Michaelson, Principal Investigator — Associate Professor, Department of Pathology, Harvard Medical School; Athanasios Zacharopoulos, Principal Investigator — Post-Doctoral Fellow, Hellenic Center for Marine Research; Christos Ouzounis, Principal Investigator — Director of Research, Centre for Research and Technology Hellas; Efstratios Karagiannidis, Principal Investigator — Phd Candidate, Aristotle University of Thessaloniki
Locations (1):
- AHEPA University Hospital, Thessaloniki, Greece

REFERENCES:
- [Background] Sianos G, Papafaklis MI, Daemen J, Vaina S, van Mieghem CA, van Domburg RT, Michalis LK, Serruys PW. Angiographic stent thrombosis after routine use of drug-eluting stents in ST-segment elevation myocardial infarction: the importance of thrombus burden. J Am Coll Cardiol. 2007 Aug 14;50(7):573-83. doi: 10.1016/j.jacc.2007.04.059. Epub 2007 Jul 30. PMID 17692740
- [Background] Ibanez B, James S, Agewall S, Antunes MJ, Bucciarelli-Ducci C, Bueno H, Caforio ALP, Crea F, Goudevenos JA, Halvorsen S, Hindricks G, Kastrati A, Lenzen MJ, Prescott E, Roffi M, Valgimigli M, Varenhorst C, Vranckx P, Widimsky P; ESC Scientific Document Group. 2017 ESC Guidelines for the management of acute myocardial infarction in patients presenting with ST-segment elevation: The Task Force for the management of acute myocardial infarction in patients presenting with ST-segment elevation of the European Society of Cardiology (ESC). Eur Heart J. 2018 Jan 7;39(2):119-177. doi: 10.1093/eurheartj/ehx393. No abstract available. PMID 28886621
- [Background] Grover SP, Saha P, Jenkins J, Mukkavilli A, Lyons OT, Patel AS, Sunassee K, Modarai B, Smith A. Quantification of experimental venous thrombus resolution by longitudinal nanogold-enhanced micro-computed tomography. Thromb Res. 2015 Dec;136(6):1285-90. doi: 10.1016/j.thromres.2015.10.006. Epub 2015 Oct 9. PMID 26489729
- [Background] Vorpahl M, Foerst JR, Kelm M, Kaplan AV, Virmani R, Ball T. The complementary role of microCT and histopathology in characterizing the natural history of stented arteries. Expert Rev Cardiovasc Ther. 2011 Jul;9(7):939-48. doi: 10.1586/erc.11.81. PMID 21809975
- [Background] Chen X, Ba Y, Ma L, Cai X, Yin Y, Wang K, Guo J, Zhang Y, Chen J, Guo X, Li Q, Li X, Wang W, Zhang Y, Wang J, Jiang X, Xiang Y, Xu C, Zheng P, Zhang J, Li R, Zhang H, Shang X, Gong T, Ning G, Wang J, Zen K, Zhang J, Zhang CY. Characterization of microRNAs in serum: a novel class of biomarkers for diagnosis of cancer and other diseases. Cell Res. 2008 Oct;18(10):997-1006. doi: 10.1038/cr.2008.282. PMID 18766170
- [Background] Navickas R, Gal D, Laucevicius A, Taparauskaite A, Zdanyte M, Holvoet P. Identifying circulating microRNAs as biomarkers of cardiovascular disease: a systematic review. Cardiovasc Res. 2016 Sep;111(4):322-37. doi: 10.1093/cvr/cvw174. Epub 2016 Jun 29. PMID 27357636